CLINICAL TRIAL: NCT06482372
Title: Effects of Repetitive Transcranial Magnetic Stimulation Combined With Mirror Therapy on Upper Limb Function in Patients With Stroke: a Pilot Study
Brief Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (1055)112A-46
Record Dates: First submitted 2024-03-17; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Mirror Therapy; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS + mirror therapy + traditional OT (Experimental): Patient would receive treatment three time per week, including individualized rTMS, and following mirror therapy and traditional occupational therapy.
  Interventions: Device: transcranial magnetic stimulation
- rTMS + traditional OT (Active Comparator): Patient would receive treatment three time per week, including individualized rTMS and following traditional occupational therapy.
  Interventions: Device: transcranial magnetic stimulation
- sham rTMS + traditional OT (Placebo Comparator): Patient would receive treatment three time per week, including sham rTMS and following traditional occupational therapy.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — repetitive transcranial magnetic stimulation at both cerebral hemisphere
  Other Names: mirror therapy

SUMMARY:
Stroke patients often have long-term upper limb dysfunction. Currently, there is still no specific clinical treatment for nerve damage. After acute treatments of stroke, patients' motor ability can only improve by spontaneous recovery of brain and rehabilitation treatment.

Transcranial magnetic stimulation uses a magnetic field pulse generated by a coil outside the skull to pass through the skull. It uses the principle that magnetic electricity can generate currents, which activates nearby brain areas or changing the relationship between the left and right brains. Transcranial magnetic stimulation is a non-invasive, safe treatment.

Mirror therapy is an emerging rehabilitation method in recent years. As mirror therapy, therapists ask the patient to place the affected hand behind the mirror while looking at the image reflected by the unaffected upper limb. During mirror therapy, patients have to perform upper limb activities and imagine that the affected upper limb is performing the same action.

As mentioned above, transcranial magnetic stimulation and mirror therapy improve the recovery of stroke patients by two different ways. Currently, there are no studies that combine these two treatments. Therefore, our study hopes to initially explore the efficacy of transcranial magnetic stimulation and the efficacy of transcranial magnetic stimulation combined with mirror therapy.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 month after stroke
* manual muscle strength < 5

Exclusion Criteria:

* history of epilepsy
* has other central nervous system diseases
* has electric medication pump
* has implant at inner ear

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) - upper extremity | week 0, week 6, week 12
  FMA would be recorded for evaluate patients' motor function of hand.
Nine-hole peg test | week 0, week 6, week 12
  Nine-hole peg test would be used to measure finger dexterity.
Action research arm test | week 0, week 6, week 12
  Action research arm test would be used to assess upper extremity performance including coordination, dexterity and functioning.
Box and block test | week 0, week 6, week 12
  Box and block test would be used to assess unilateral gross manual dexterity.
Functional independence measurement | week 0, week 6, week 12
  Functional independence measurement would be recorded to assess a patient's level of disability as well as a change in patient status in response to rehabilitation or medical intervention.

IPD SHARING:
Plan to Share IPD: Undecided